CLINICAL TRIAL: NCT03829839
Title: Common and Dissociable Effects of Oxytocin and Lorazepam on the Neurocircuitry of Fear - an Ultra-high Field Imaging Study
Brief Title: Effects of Oxytocin and Lorazepam on Fear-related Intra-amygdalar Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Vice Chair of the Department of Psychiatry and Chair of the Medical Psychology Division, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: LOXY
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Oxytocin, Lorazepam, Anti-Anxiety Agents, Physiological Effects of Drugs
Keywords: Amygdala, anxiety, benzodiazepines, fear, fMRI, lorazepam, oxytocin, 7 Tesla
MeSH Terms: conditions — Anxiety Disorders | interventions — Oxytocin; Lorazepam; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin or PLC (Active Comparator): Single dose of intranasal oxytocin (24 international units) or PLC.
  Interventions: Drug: Oxytocin; Drug: Placebo nasalspray
- Lorazepam or PLC (Active Comparator): Single dose of lorazepam (1mg) or PLC
  Interventions: Drug: Lorazepam 1 mg; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Oxytocin — Intranasal administration, 24 international units (IU) oxytocin
  Other Names: syntocinon
  Arms: Oxytocin or PLC
Drug: Lorazepam 1 mg — Oral administration of 1mg lorazepam
  Other Names: Tavor
  Arms: Lorazepam or PLC
Drug: Placebo nasalspray — The placebo nasalspray contain identical ingredients except for the active agent itself.
  Arms: Oxytocin or PLC
Drug: Placebo Oral Tablet — The placebo pill contain identical ingredients except for the active agent itself.
  Arms: Lorazepam or PLC

SUMMARY:
High-potency benzodiazepines have strong anxiolytic effects accompanied by significant adverse effects including impaired cognitive function, drowsiness, dizziness and impaired motoric abilities. Importantly, the long-term use of benzodiazepines may produce dependence and withdrawal. Therefore, there is considerable scientific and public interest in identifying new anxiolytic agents.

The hypothalamic peptide oxytocin (OXT) has anxiolytic effects both in healthy participants and patients with anxiety disorders by decreasing fear-associated amygdala activity. However, so far no human study has directly compared the underlying anxiolytic mechanisms of OXT and established anxiolytic agents on amygdala activity. Importantly, the amygdala is not a homogenous structure but rather consists of several subdivisions with structural and functional differences.

Therefore, the rationale of the present project is to determine the effects of intranasal OXT and the high-potency benzodiazepine lorazepam on fear-associated responses in intra-amygdalar subregions.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers
* right-handed

Exclusion Criteria:

* Current or past psychiatric illness
* Current or past physical illness
* Psychoactive medication
* Sedative medication
* MRI contraindication (e.g. metal in body, claustrophobia)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Neural responses to emotional faces in the amygdala subregions | Neural activations with be measured with 7 Tesla fMRI in an emotional face matching task that lasts 20 mins
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli. The investigators specifically plan to investigate amygdala subregion responses to emotional faces.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://renehurlemann.squarespace.com/welcome/